CLINICAL TRIAL: NCT02497235
Title: An Open-Label, Positron Emission Tomography, Phase 1 Study With [18F]MNI-792 to Determine Cholesterol 24S-Hydroxylase Target Occupancy of TAK-935 After Single-Dose Oral Administration in Healthy Subjects.
Brief Title: A Phase 1 Positron Emission Tomography Study to Measure Cholesterol 24S-Hydroxylase Target Occupancy of TAK-935
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAK-935_1003; U1111-1170-0452 (Registry Identifier: WHO)
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Epilepsy, Molecular Mechanisms of Pharmalogical Action, Protective Agents
Keywords: Drug therapy, Positron Emission Tomography, Brain enzyme occupancy, Cholesterol 24S-hydroxylase, CH24H
MeSH Terms: conditions — Epilepsy | interventions — Product Labeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-935 (Experimental): A single dose of TAK-935 600 milligram (mg), oral solution on Day 1 as a starting dose and up to 370 megabecquerel (MBq) (10 millicurie [mCi]) of [18F]MNI-792 with a mass of up to 5 microgram (mcg), injection intravenously (IV), prior to each PET imaging at Baseline, 45 minutes and 10 hours post-TAK-935 dose. Subsequent dose of TAK-935 oral solution and timing of PET imaging will be based on safety, tolerability and occupancy data from previous level participants.
  Interventions: Drug: TAK-935; Drug: [18F]MNI-792 (tracer)

INTERVENTIONS:
Drug: TAK-935 — TAK-935 oral solution.
Drug: [18F]MNI-792 (tracer) — [18F]MNI-792 injection.

SUMMARY:
The purpose of this study is to determine the brain cholesterol 24S-hydroxylase (CH24H) enzyme occupancy of TAK-935 after single oral dose in healthy participants using the positron emission tomography (PET) ligand [18F]MNI-792 and PET imaging and to determine the relationship of occupancy to TAK-935 exposure.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-935. TAK-935 is being tested to examine the degree and duration of brain CH24H enzyme occupancy/target engagement as a function of TAK-935 plasma concentration in order to guide dosing and schedule for future clinical trials with TAK-935. This study will utilize the PET ligand [18F]MNI-792 to evaluate the brain CH24H occupancy of TAK-935 after single dose oral administration in healthy adult participants. The study will evaluate up to 16 participants. The first 2 participants will take TAK-935 600 mg oral solution and undergo PET imaging using tracer [18F]MNI-792 up to 5 mcg (up to 370 MBq), injection, intravenously prior to each PET scan at Baseline, 45 minutes and 10 hours post-TAK-935 dose. TAK-935 dose and timing of post-dose scans for subsequent participants will be based on the data from the previous participants. This single-center trial will be conducted in the United States. The overall time to participate in this study is up to 55 days. Participants will make 4 visits to the clinic, including 2 confinement periods to the clinic for PET imaging. Participants will be contacted by phone on Day 28 for follow-up safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, is capable of understanding and complying with protocol requirements.
2. Signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures including requesting that a participant fast for any laboratory evaluations.
3. Is a healthy male or female and aged 19 to 55 years, inclusive, at the time of informed consent and first study medication dose.
4. Weighs at least 45 kilogram (kg) and has a body mass index (BMI) from 18.0 to 30.0 kilogram per square meter (kg/m^2), inclusive at Screening.
5. A female of non-bearing potential (example post-menopausal by history; or history of hysterectomy, bilateral salpingectomy, or oophorectomy).

Exclusion Criteria:

1. Have a known history or evidence of a clinically significant disorder (including neurologic and psychiatric), or disease that in the opinion of the study investigator would pose a risk to the participant safety or interfere with the study evaluation, procedures or completion.
2. Contraindication to magnetic resonance imaging (MRI) based on the standard MRI radiography screening questionnaire.
3. Had exposure to any radiation greater than (>) 15 millisievert (mSv)/year (example, occupational or radiation therapy) within the previous year prior to Baseline imaging.
4. Has a known hypersensitivity to any component of the formulation of TAK-935 or related compounds, or to [18F]MNI-792 or to any of its components.
5. Clinically significant abnormal findings on brain MRI scan or findings on brain MRI that may interfere with the interpretation of the PET imaging.
6. Use of any over-the-counter, herbal, or prescription medications or supplements within 30 days prior to baseline imaging.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- New Haven, Connecticut, United States

REFERENCES:
- [Derived] Constantinescu CC, Brown T, Wang S, Yin W, Barret O, Jennings D, Tauscher J. Clinical Characterization of [18F]T-008, a Cholesterol 24-Hydroxylase PET Ligand: Dosimetry, Kinetic Modeling, Variability, and Soticlestat Occupancy. J Nucl Med. 2023 Dec 1;64(12):1972-1979. doi: 10.2967/jnumed.123.265912. PMID 37770111

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 01 July 2015 to 04 January 2016.
Pre-assignment Details: Healthy participants received up to 370 megabecquerel (MBq) (10 millicurie [mCi]) of [18F]MNI-792 with a mass of up to 5 microgram (mcg) at baseline and were enrolled to 1 of 5 treatment groups: TAK-935 50 milligram (mg), 100 mg, 200 mg, 300 mg, and 600 mg.
Groups:
- TAK-935 50 mg: TAK-935 50 mg, solution, orally, once on Day 1 and up to 370 MBq (10 mCi) of [18F]MNI-792 with a mass of up to 5 mcg, injection, intravenously, prior to PET imaging at 2 hours and 24 hours post-TAK-935 dose.
- TAK-935 100 mg: TAK-935 100 mg, solution, orally, once on Day 1 and up to 370 MBq (10mCi) of [18F]MNI-792 with a mass of up to 5 mcg, injection, intravenously, prior to PET imaging at Baseline, 2 hours and 24 hours post-TAK-935 dose.
- TAK-935 200 mg: TAK-935 200 mg, solution, orally, once on Day 1 and up to 370 MBq (10mCi) of [18F]MNI-792 with a mass of up to 5 mcg, injection, intravenously, prior to PET imaging at Baseline, 2 hours and 24 hours post-TAK-935 dose.
- TAK-935 300 mg: TAK-935 300 mg, solution, orally, once on Day 1 and up to 370 MBq (10mCi) of [18F]MNI-792 with a mass of up to 5 mcg, injection, intravenously, prior to PET imaging at Baseline, 2 hours and 24 hours post-TAK-935 dose.
- TAK-935 600 mg: TAK-935 600 mg, solution, orally, once on Day 1 and up to 370 MBq (10mCi) of [18F]MNI-792 with a mass of up to 5 mcg, injection, intravenously, prior to first PET imaging at Baseline, 45 minutes and 10 hours post-TAK-935 dose for the first 2 enrolled participants and at Baseline, 2 hours and 24 hours post-TAK-935 dose for the participant enrolled later.
Period: Overall Study
Arm/Group | TAK-935 50 mg | TAK-935 100 mg | TAK-935 200 mg | TAK-935 300 mg | TAK-935 600 mg
Started | 2 | 2 | 2 | 2 | 3
Completed | 2 | 2 | 2 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were enrolled and received investigational drug ([18F]MNI-792 or TAK-935).
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-935 50 mg | TAK-935 100 mg | TAK-935 200 mg | TAK-935 300 mg | TAK-935 600 mg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (7.07) | 25.5 (2.12) | 42.0 (2.83) | 48.5 (2.12) | 36.7 (6.11) | 38.4 (8.48)
Sex/Gender, Customized [Number; unit: participants]
  Male | 2 | 2 | 2 | 2 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 2 | 2 | 3 | 11
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 1 | 4
  Not Hispanic or Latino | 1 | 0 | 2 | 2 | 2 | 7
Race [Number; unit: participants]
  Black or African American | 2 | 1 | 2 | 0 | 1 | 6
  White | 0 | 1 | 0 | 2 | 2 | 5
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 171.5 (4.95) | 181.5 (3.54) | 177.0 (4.24) | 180.0 (0.00) | 183.0 (16.09) | 179.0 (8.69)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 86.05 (7.283) | 93.60 (10.748) | 79.40 (12.869) | 87.05 (5.162) | 84.83 (23.692) | 86.06 (13.009)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 29.22 (0.789) | 28.37 (2.157) | 25.46 (5.327) | 26.87 (1.593) | 24.95 (4.275) | 26.79 (3.212)

OUTCOME MEASURES:

1. Primary Outcome: Cholesterol 24S-Hydroxylase (CH24H) Brain Enzyme Occupancy as a Function of TAK-935 Plasma Concentration at 45 Minutes Post-TAK-935 Dose
Description: CH24H brain enzyme occupancy was obtained by graphical analysis of global occupancy plot. Global occupancy plot was calculated as: total volume of distribution [VT] (Baseline) - VT (Day 1) = Occupancy (Day 1) * (VT [Baseline] - non-displaceable volume of distribution [VND]), where VT (Baseline) and VT (Day 1) are the total distribution volumes obtained at Baseline and after TAK-935 administration, respectively and VND is the non-displaceable volume of distribution. The occupancy is determined as the slope of the linear regression of the plot, and the VND as the x-intercept. Data was reported only for TAK-935 600 mg because only first two participants were analyzed at 45 minutes post-TAK-935 dose.
Time Frame: 45 minutes post-TAK-935 dose
Population: PET target occupancy set where 45 minutes post-TAK-935-dose assessment were available. PET target occupancy set included all participants who received study drug (TAK-935) and had a technically adequate Baseline PET scan and at least 1 technically adequate post-TAK-935 dose PET scan.
Measure: Number; unit: percentage of occupancy
Groups:
- TAK-935 600 mg: TAK-935 600 mg, solution, orally, once on Day 1 and up to 370 MBq (10mCi) of [18F]MNI-792 with a mass of up to 5 mcg, injection, intravenously, prior to first PET imaging at Baseline, 45 minutes and 10 hours post-TAK-935 dose for the first 2 enrolled participants.
Arm/Group | TAK-935 600 mg
Number analyzed (Participants) | 2
percentage of occupancy
  Participant 1 | NA — Data was not reported because post dose imaging data was not quantifiable.
  Participant 2 | 98
  Participant 3 | NA — Data was not reported because only two participants were analyzed at 45 minutes post-TAK-935.

2. Primary Outcome: CH24H Brain Enzyme Occupancy as a Function of TAK-935 Plasma Concentration at 2 Hours Post-TAK-935 Dose
Description: CH24H brain enzyme occupancy was obtained by graphical analysis of global occupancy plot. Global occupancy plot was calculated as: VT (Baseline) - VT (Day 1) = Occupancy (Day 1) * (VT [Baseline] - VND), where VT (Baseline) and VT (Day 1) are the total distribution volumes obtained at Baseline and after TAK-935 administration, respectively and VND is the non-displaceable volume of distribution. The occupancy is determined as the slope of the linear regression of the plot, and the VND as the x-intercept.
Time Frame: 2 hours post-TAK-935 dose
Population: PET target occupancy set where 2 hour post-TAK-935-dose assessment were available. PET target occupancy set included all participants who received study drug (TAK-935) and had a technically adequate Baseline PET scan and at least 1 technically adequate post-TAK-935 dose PET scan.
Measure: Number; unit: percentage of occupancy
Groups:
- TAK-935 600 mg: TAK-935 600 mg, solution, orally, once on Day 1 and up to 370 MBq (10mCi) of [18F]MNI-792 with a mass of up to 5 mcg, injection, intravenously, prior to first PET imaging at Baseline, 2 hours and 24 hours post-TAK-935 dose for the participant enrolled later.
Arm/Group | TAK-935 50 mg | TAK-935 100 mg | TAK-935 200 mg | TAK-935 300 mg | TAK-935 600 mg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 1
percentage of occupancy
  Participant 1 | 70 | 79 | 96 | 91 | NA — Data not reported because participant was not imaged at 2 hours post-TAK-935 600 mg dose.
  Participant 2 | 64 | 85 | 89 | 89 | NA — Data not reported because participant was not imaged at 2 hours post-TAK-935 600 mg dose.
  Participant 3 | NA — Data was not reported because only two participants were analyzed at 2 hour post-TAK-935 dose. | NA — Data was not reported because only two participants were analyzed at 2 hour post-TAK-935 dose. | NA — Data was not reported because only two participants were analyzed at 2 hour post-TAK-935 dose. | NA — Data was not reported because only two participants were analyzed at 2 hour post-TAK-935 dose. | 96

3. Primary Outcome: CH24H Brain Enzyme Occupancy as a Function of TAK-935 Plasma Concentration at 10 Hours Post-TAK-935 Dose
Description: CH24H brain enzyme occupancy was obtained by graphical analysis of global occupancy plot. Global occupancy plot was calculated as: VT (Baseline) - VT (Day 1) = Occupancy (Day 1) * (VT [Baseline] - VND), where VT (Baseline) and VT (Day 1) are the total distribution volumes obtained at Baseline and after TAK-935 administration, respectively and VND is the non-displaceable volume of distribution. The occupancy is determined as the slope of the linear regression of the plot, and the VND as the x-intercept. Data was reported only for TAK-935 600 mg because only first two participants were analyzed at 10 hour post-TAK-935 dose.
Time Frame: 10 hours post-TAK-935 dose
Population: PET target occupancy set where 10 hour post-TAK-935-dose assessment were available. PET target occupancy set included all participants who received study drug (TAK-935) and had a technically adequate Baseline PET scan and at least 1 technically adequate post-TAK-935 dose PET scan.
Measure: Number; unit: percentage of occupancy
Arm/Group | TAK-935 600 mg
Number analyzed (Participants) | 2
percentage of occupancy
  Participant 1 | 92
  Participant 2 | 87
  Participant 3 | NA — Data not reported because Participant 3 was not imaged at 10 hours post-TAK-935 600 mg dose.

4. Primary Outcome: CH24H Brain Enzyme Occupancy as a Function of TAK-935 Plasma Concentration at 24 Hours Post-TAK-935 Dose
Description: as for outcome 2
Time Frame: 24 hours post-TAK-935 dose
Population: PET target occupancy set where 24 hour post-TAK-935-dose assessment were available. PET target occupancy set included all participants who received study drug (TAK-935) and had a technically adequate Baseline PET scan and at least 1 technically adequate post-TAK-935 dose PET scan.
Measure: Number; unit: percentage of occupancy
Arm/Group | TAK-935 50 mg | TAK-935 100 mg | TAK-935 200 mg | TAK-935 300 mg | TAK-935 600 mg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 1
percentage of occupancy
  Participant 1 | 22 | 13 | 79 | 46 | NA — Data not reported because participant was not imaged at 24 hours post-TAK-935 600 mg dose.
  Participant 2 | 11 | NA — Data was not reported due to non-availability of blood data for second dose scan. | 47 | 27 | NA — Data not reported because participant was not imaged at 24 hours post-TAK-935 600 mg dose.
  Participant 3 | NA — Data was not reported because only two participants were analyzed at 24 hour post-TAK-935 dose. | NA — Data was not reported because only two participants were analyzed at 24 hour post-TAK-935 dose. | NA — Data was not reported because only two participants were analyzed at 24 hour post-TAK-935 dose. | NA — Data was not reported because only two participants were analyzed at 24 hour post-TAK-935 dose. | 52

5. Secondary Outcome: Plasma Concentration of TAK-935 During Post-TAK-935 Dosing PET Scan Periods
Time Frame: At time 0 (just after tracer injection), 1 hour after tracer injection and 2 hours after tracer injection for each post-TAK-935 dosing PET scan period
Population: Pharmacokinetic (PK) set included all participants who received TAK-935 and had at least 1 measurable plasma concentration for either TAK-935 or its M-1 metabolite. Data was reported for Participant 1 and 2 of each of TAK-935 50, 100, 200, and 300 mg arms and Participant 1, 2, and 3 of TAK-935 600 mg arm.
Measure: Number; unit: nanogram per milliliter (ng/mL)
Arm/Group | TAK-935 50 mg | TAK-935 100 mg | TAK-935 200 mg | TAK-935 300 mg | TAK-935 600 mg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3
nanogram per milliliter (ng/mL)
  Participant 1: PET Scan 1: pre-tracer dose | 9.16 | 11.3 | 158 | 56.2 | 6.83
  Participant 1: PET Scan 1: 1 hour post-tracer dose | 3.79 | 5.02 | 72.7 | 19.4 | 200
  Participant 1:PET Scan 1: 2 hours post-tracer dose | 2.98 | 2.45 | 30.3 | 12.9 | 379
  Participant 1: PET Scan 2: pre-tracer dose | NA — Data could not be analyzed because data was below the limit of quantitation. | NA — Data could not be analyzed because data was below the limit of quantitation. | 14.2 | NA — Data could not be analyzed because data was below the limit of quantitation. | 22.3
  Participant 1:PET Scan 2: 1 hour post-tracer dose | NA — Data could not be analyzed because data was below the limit of quantitation. | NA — Data could not be analyzed because data was below the limit of quantitation. | 9.16 | NA — Data could not be analyzed because data was below the limit of quantitation. | 16
  Participant 1:PET Scan 2:2 hours post-tracer dose | NA — Data could not be analyzed because data was below the limit of quantitation. | NA — Data could not be analyzed because data was below the limit of quantitation. | 8.08 | NA — Data could not be analyzed because data was below the limit of quantitation. | 14.4
  Participant 2: PET Scan 1: pre-tracer dose | 6.92 | 23.9 | 34.8 | 50.9 | 569
  Participant 2: PET Scan 1: 1 hour post-tracer dose | 2.97 | 12.3 | 16.8 | 15.7 | 257
  Participant 2:PET Scan 1: 2 hours post-tracer dose | 1.95 | 6.46 | 7.52 | 14.6 | 90.8
  Participant 2: PET Scan 2: pre-tracer dose | NA — Data could not be analyzed because data was below the limit of quantitation. | 1.83 | NA — Data could not be analyzed because data was below the limit of quantitation. | NA — Data could not be analyzed because data was below the limit of quantitation. | 7.99
  Participant 2:PET Scan 2: 1 hour post-tracer dose | NA — Data could not be analyzed because data was below the limit of quantitation. | 1.28 | NA — Data could not be analyzed because data was below the limit of quantitation. | NA — Data could not be analyzed because data was below the limit of quantitation. | 6.27
  Participant 2:PET Scan 2:2 hours post-tracer dose | NA — Data could not be analyzed because data was below the limit of quantitation. | NA — Data could not be analyzed because data was below the limit of quantitation. | NA — Data could not be analyzed because data was below the limit of quantitation. | NA — Data could not be analyzed because data was below the limit of quantitation. | 5.12
  Participant 3: PET Scan 1: pre-tracer dose | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | 589
  Participant 3: PET Scan 1: 1 hour post-tracer dose | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | 236
  Participant 3:PET Scan 1: 2 hours post-tracer dose | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | 155
  Participant 3: PET Scan 2: pre-tracer dose | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | 3.04
  Participant 3: PET Scan 2: 1 hour post-tracer dose | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | 2.58
  Participant 3:PET Scan 2: 2 hours post-tracer dose | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | 2.24

6. Secondary Outcome: Percent Change From Baseline in the AUEC24 for Plasma 24S Hydroxycholesterol (24HC)
Description: Percent change was calculated as = [(Postdose AUEC24(2) - Baseline AUEC24(2))/Baseline AUEC24(2)]*100 percent.
Time Frame: Baseline (Day -1): 1 hour and at multiple timepoints (up to 12 hours) post check in and Day 1: pre-dose and at multiple timepoints (up to 24 hours) post-TAK-935 dose
Population: PK set included all participants who received TAK-935 and had at least 1 measurable plasma concentration for either TAK-935 or its M-1 metabolite. Data was reported for Participant 1 and 2 of each of TAK-935 50, 100, 200, and 300 mg arms and Participant 1, 2, and 3 of TAK-935 600 mg arm.
Measure: Number; unit: percent change
Arm/Group | TAK-935 50 mg | TAK-935 100 mg | TAK-935 200 mg | TAK-935 300 mg | TAK-935 600 mg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3
percent change
  Participant 1 | -6.79 | -14.82 | -10.50 | -12.41 | -7.23
  Participant 2 | -13.38 | -15.04 | -9.30 | -18.55 | -12.79
  Participant 3 | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | -6.81

ADVERSE EVENTS:
Time Frame: Baseline up to Day 28
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Adverse events were summarized separately for Baseline period and TAK-935 dosing groups.
Groups:
- Baseline [18F]MNI-792: [18F]MNI-792 up to 370 MBq (10mCi) with a mass of up to 5 mcg, injection, intravenously, prior to Positron Emission Tomography (PET) imaging at Baseline.
- TAK-935 100 mg: TAK-935 100 mg, solution, orally, once on Day 1 and up to 370 MBq (10mCi) of [18F]MNI-792 with a mass of up to 5 mcg, injection, intravenously, prior to PET imaging at 2 hours and 24 hours post-TAK-935 dose.
- TAK-935 200 mg: TAK-935 200 mg, solution, orally, once on Day 1 and up to 370 MBq (10mCi) of [18F]MNI-792 with a mass of up to 5 mcg, injection, intravenously, prior to PET imaging at 2 hours and 24 hours post-TAK-935 dose.
- TAK-935 300 mg: TAK-935 300 mg, solution, orally, once on Day 1 and up to 370 MBq (10mCi) of [18F]MNI-792 with a mass of up to 5 mcg, injection, intravenously, prior to PET imaging at 2 hours and 24 hours post-TAK-935 dose.
- TAK-935 600 mg: TAK-935 600 mg, solution, orally, once on Day 1 and up to 370 MBq (10mCi) of [18F]MNI-792 with a mass of up to 5 mcg, injection, intravenously, prior to first PET imaging at 45 minutes and 10 hours post-TAK-935 dose for the first 2 enrolled participants and at 2 hours and 24 hours post-TAK-935 dose for the participant enrolled later.
Arm/Group | Baseline [18F]MNI-792 | TAK-935 50 mg | TAK-935 100 mg | TAK-935 200 mg | TAK-935 300 mg | TAK-935 600 mg
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/2 | 0/2 | 0/2 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 1/11 | 1/2 | 1/2 | 1/2 | 1/2 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Baseline [18F]MNI-792 (N=11) | TAK-935 50 mg (N=2) | TAK-935 100 mg (N=2) | TAK-935 200 mg (N=2) | TAK-935 300 mg (N=2) | TAK-935 600 mg (N=3)
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0/1 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.